CLINICAL TRIAL: NCT05411042
Title: Benefits of Digital Dance Game Participation by Older Adults on Brain Gray Matter Volume, Physical Function, Cognitive Performance, and Quality of Life: a Randomized Controlled Trial.
Brief Title: Benefits of Digital Dance Game by Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YM108123F_D
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2020-06

CONDITIONS: Aged
Keywords: Digital dance game; older adults; Brain gray matter volume; cognitive performance

STUDY DESIGN:
Intervention Model Description: The intervention group and control group were randomly allocated (1:1) with no stratification. The intervention group received the dance somatosensory videogame (DSG) training program at the community health center, which consisted of two 30-minute sessions per week for 6 months. The control group were provided with health education for healthy aging and were followed by telephone survey for their daily activities every month during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group intervened a dance somatosensory game (DSG), DANZ BASE developed by International Games System Company, at the Xinzhuang health center, which is a local bureau with outpatient clinic. The participants in experimental group played twice a week, each time requiring at least lasting 30 minutes, for half of a year.
  Interventions: Device: Dance somatosensory game
- Control group (No Intervention): The control group only performed routine data collection; the research assistant asked the subjects about their usual activities by telephone every month to understand their physical activity in this half of the year.

INTERVENTIONS:
Device: Dance somatosensory game — dance somatosensory game (DSG), DANZ BASE developed by International Games System Company
  Arms: Intervention group

SUMMARY:
This study aims to examine the clinical efficacy of dancing somatosensory videogames in improving physical health, cognitive performance, happiness, laboratory biomarkers, and structural brain imaging (magnetic resonance imaging, MRI) by a randomized controlled trial design, and hopefully to expand the scope of healthy aging intervention activities with strong scientific evidence.

DETAILED DESCRIPTION:
This randomized controlled trial followed the CONSORT guidelines to compare the clinical efficacy of the intervention group with the control group. The intervention group and control group were randomly allocated (1:1) with no stratification. The intervention group received the dance somatosensory videogame (DSG) training program at the community health center, which consisted of two 30-minute sessions per week for 6 months. The control group were provided with health education for healthy aging and were followed by telephone survey for their daily activities every month during the study period.

The primary outcome of the trial was changes of gray matter volume of the brain done by 3T brain magnetic resonance imaging during the study period. The secondary outcomes included cognitive performance, quality of life, physical activities, resilience, and demoralization. For all outcome variables, the measurements at the baseline and 6-month follow-up were examined by a random intercept and a fixed slope, and the effect of the intervention was estimated by using the Generalized Estimating Equation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 55 years old.
2. More than 6 years of formal education.
3. Can communicate in Mandarin and Taiwanese.
4. Can accept MRI examination without claustrophobia.
5. Can understand the research process, meet the requirements of the research, and can sign the consent form and participate in the subject.

Exclusion Criteria:

1. Have engaged in any video dancing games in the past three months.
2. Engaged in video dancing games more than three times per year in the past three years.

Ages: 55 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Change in MRI study | from baseline to 6 months
  Change in MRI study from baseline to 6 months in the intervention group.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | from baseline to 6 months
  Cognitive function measure by MoCA , which comprise a 30-question test.Score range: 0-30, and a score of 26 and higher is considered normal.
EuroQol instrument (EQ-5D) | from baseline to 6 months
  Quality of life measure by EQ-5D, which include five questions on mobility, self care, pain, usual activities, and psychological status.There are three level of the answers for each question, the maximum score of 1 refers to the best condition without problem, and higher scores refers more severe of the issue. Moreover, the visual analogue scale (VAS) which from 0-100, higher score indicating better health status.
International Physical Activity Questionnaire (IPAQ) | from baseline to 6 months
  Physical activity measured by IPAQ, indicates that spent being physically active within the prior 7 days.There are no established thresholds for presenting MET-minutes, the IPAQ Research Committee proposes that reported as comparisons of median values and interquartile ranges for different populations.
Brief Resilience Scale (BRS) | from baseline to 6 months
  Resilience measured by BRS to assess ability to bounce back or recover from stress and adversity. Score range: 6-30, and higher scores refers to higher level of resilience.
Demoralization Scale-Mandarin Version (DS-MV) | from baseline to 6 months
  Demoralization measure by DS-MV, comprised 24 items and each rated on a five-point Likert scale.Score range: 0-96, and cut-off point score ≥30 was considered to identified demoralization.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, M.D., PhD, Study Director — Aging and Health Research Center, National Yang-Ming University
Locations (1):
- Center for Geriatrics and Gerontology, Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tung HH, Kuo CY, Lee PL, Chang CW, Chou KH, Lin CP, Chen LK. Efficacy of Digital Dance on Brain Imagery, Cognition, and Health: Randomized Controlled Trial. J Med Internet Res. 2024 Jul 30;26:e57694. doi: 10.2196/57694. PMID 39078687